CLINICAL TRIAL: NCT02719964
Title: Rehabilitation of Visual Attention Following mTBI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: United States Naval Medical Center, San Diego (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NMCSD.2015.0049
Record Dates: First submitted 2016-03-21; First posted 2016-03-25 (Estimated); Last update posted 2019-03-13 (Actual); Status verified 2019-03

CONDITIONS: Traumatic Brain Injury
Keywords: Cognitive Training; Traumatic Brain Injury; Video Games
MeSH Terms: conditions — Brain Injuries, Traumatic

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (4):
- A: UCR Games→SP-Directed Therapy (Experimental): Participants in Arm A will first participate in Visual Attention Program (UCR Games) followed by Speech Pathologist-Directed Therapy with assessment sessions prior to and following each treatment intervention.
  Interventions: Other: Visual Attention Program (UCR Games); Other: Speech Pathologist-Directed Therapy
- B: Lumosity→SP-Directed Therapy (Experimental): Participants in Arm B will first participate in General Cognitive Rehabilitation Games (Lumosity) followed by Speech Pathologist-Directed Therapy with assessment sessions prior to and following each treatment intervention.
  Interventions: Other: Speech Pathologist-Directed Therapy; Other: General Cognitive Rehabilitation Games (Lumosity)
- C: SP-Directed Therapy→UCR Games (Experimental): Participants in Arm C will first participate in Speech Pathologist-Directed Therapy followed by Visual Attention Program (UCR Games) with assessment sessions prior to and following each treatment intervention.
  Interventions: Other: Visual Attention Program (UCR Games); Other: Speech Pathologist-Directed Therapy
- D: SP-Directed Therapy→Lumosity (Experimental): Participants in Arm D will first participate in Speech Pathologist-Directed Therapy followed by General Cognitive Rehabilitation Games (Lumosity) with assessment sessions prior to and following each treatment intervention.
  Interventions: Other: Speech Pathologist-Directed Therapy; Other: General Cognitive Rehabilitation Games (Lumosity)

INTERVENTIONS:
Other: Visual Attention Program (UCR Games) — This program is an individual-directed computerized cognitive rehabilitation program based on perceptual learning approaches to enhance visual attention. Training incorporates a diverse set of stimuli, optimized stimulus presentation, multisensory facilitation, and consistently reinforcing training stimuli. This will be completed in a group setting with an instructor available to facilitate questions.
  Arms: A: UCR Games→SP-Directed Therapy; C: SP-Directed Therapy→UCR Games
Other: Speech Pathologist-Directed Therapy — This is a speech pathologist-directed arm and will provide a traditional clinician-directed individualized cognitive rehabilitation program. Cognitive treatment is a systematic, functionally oriented program of therapeutic activities that focuses on strengthening previously learned patterns of behavior, establishing new patterns through use of internal and external compensatory cognitive strategies, and enabling the individual to adapt to the changes in his or her revised approaches to cognitive functioning. Increased performance success is reinforced through repetition, errorless learning, and gradually increasing task stimuli and complexity in a structured systematic approach.
Other: General Cognitive Rehabilitation Games (Lumosity) — Lumosity is a commercially available computerized program purported to enhance cognitive functioning through a variety of computerized programs that utilize various cognitive abilities.
  Arms: B: Lumosity→SP-Directed Therapy; D: SP-Directed Therapy→Lumosity

SUMMARY:
The objective of this proposal is to evaluate the effectiveness of rehabilitation for visual attention deficits in U.S. military service members across three programs: Visual Attention and Working Memory Programs (UCR Games), Speech Pathologist-Directed Treatment, and General Cognitive Rehabilitation Games (Lumosity).

In addition to the above prospective component, this study also has a retrospective component in which archival data collected from routine clinical care will be examined for analysis. The investigators hope to gain a better understanding of the unique and cumulative influence different cognitive rehabilitation programs have on improving attention complaints in mTBI.

DETAILED DESCRIPTION:
Mild traumatic brain injury (mTBI) is one of the most commonly sustained combat-related injuries. Complaints of poor attention often follow mTBI and can become chronic in some individuals. Chronic attention complaints have traditionally been treated with cognitive rehabilitation by speech pathologists. Recent research has shown that computerized programs may add additional value either independently or in conjunction with traditional therapies. Researchers at UC Riverside have already completed research showing that vision training, using the ULTIMEYES program that they created, led to improved vision both on standard assessments, such as reading eye-charts, and in real world skills, such as reading and playing baseball. This program is designed to broadly improve basic aspects of vision, such as visual acuity and contrast sensitivity, as well as high-level vision, such as attention. Furthermore, an associated memory training task (Recall The Game) shows improvements in memory tasks and transfer to skills such as fluid intelligence.

The objective of this proposal is to evaluate the effectiveness of rehabilitation for visual attention deficits in U.S. military service members across three programs:

1. Visual Attention and Memory Program (UCR Games)
2. Cognitive and Psychological Based Rehabilitation (Speech Pathologist-Directed Therapy)
3. General Cognitive Rehabilitation Games (Lumosity [2])

The investigators hope to gain a better understanding of the unique and cumulative influence of different cognitive rehabilitation programs on improving attention complaints in mTBI. This proposal contains both retrospective and prospective components.

The retrospective component consists of examining archival data from Lumosity, previously collected as part of routine clinical care. The data contain pre- and post-assessments of post-concussive symptoms, symptom frequency, and cognitive testing. The investigators expect that data analysis will reveal evidence of improvement in severity of post-concussive symptoms, in frequency of troublesome cognitive problems, and in performance on neuropsychological tests when pre- and post-assessments are compared.

The prospective component will consist of 120 service members with mTBI who have ongoing attention complaints and are more than three months post-injury. Each service member will be randomly assigned to one of four arms, differentiated only by the specific computer-based rehabilitation program used. All individuals will also be treated per current standard of care guidelines by a speech pathologist.

Each of the four arms will be comprised of 30 participants. A cognitive testing battery will be administered to each participant before and after implementation of each intervention. The cognitive testing battery form will vary based on time of administration in order to control for practice effects. Performance on the cognitive testing battery and self-report measures will be compared between and within the three arms.

This research will help the military to identify the best cognitive rehabilitation treatment program to address ongoing attention complaints following mTBI.

ELIGIBILITY:
Inclusion Criteria:

* Closed TBI
* Have sufficient information available that we can confidently classify severity as mild based on DOD/VA criteria
* Time tested post-injury > 3 months
* Ongoing attention complaints

Exclusion Criteria:

* Moderate/Severe TBI
* Penetrating TBI
* Attention Deficit Hyperactivity Disorder
* Learning Disorder
* Diagnosed medical condition that is expected to impact cognitive performance (i.e. Multiple Sclerosis, Stroke)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2016-05; Primary Completion 2020-10 (Estimated); Study Completion 2020-10 (Estimated)

PRIMARY OUTCOMES:
Post-Concussion Cognitive Symptoms | Two Months
  Comparison of performance on pre- and post-intervention neuropsychological testing battery.
Severity of Post-Concussive Symptoms | Two Months
  Comparison of self-reported symptoms on pre- and post-intervention assessment.

CONTACTS AND LOCATIONS:
Overall Officials: Brittany E Powell, MD, Principal Investigator — United States Naval Medical Center, San Diego
Locations (1):
- Naval Medical Center San Diego, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Deveau J, Ozer DJ, Seitz AR. Improved vision and on-field performance in baseball through perceptual learning. Curr Biol. 2014 Feb 17;24(4):R146-7. doi: 10.1016/j.cub.2014.01.004. No abstract available. PMID 24556432
- [Background] Lumosity. Available from: http://www.lumosity.com.
- [Background] Carey ME. Learning from traditional combat mortality and morbidity data used in the evaluation of combat medical care. Mil Med. 1987 Jan;152(1):6-13. No abstract available. PMID 3103012
- [Background] Hoge CW, McGurk D, Thomas JL, Cox AL, Engel CC, Castro CA. Mild traumatic brain injury in U.S. Soldiers returning from Iraq. N Engl J Med. 2008 Jan 31;358(5):453-63. doi: 10.1056/NEJMoa072972. Epub 2008 Jan 30. PMID 18234750
- [Background] Schneiderman AI, Braver ER, Kang HK. Understanding sequelae of injury mechanisms and mild traumatic brain injury incurred during the conflicts in Iraq and Afghanistan: persistent postconcussive symptoms and posttraumatic stress disorder. Am J Epidemiol. 2008 Jun 15;167(12):1446-52. doi: 10.1093/aje/kwn068. Epub 2008 Apr 17. PMID 18424429
- [Background] Schwab KA, Ivins B, Cramer G, Johnson W, Sluss-Tiller M, Kiley K, Lux W, Warden D. Screening for traumatic brain injury in troops returning from deployment in Afghanistan and Iraq: initial investigation of the usefulness of a short screening tool for traumatic brain injury. J Head Trauma Rehabil. 2007 Nov-Dec;22(6):377-89. doi: 10.1097/01.HTR.0000300233.98242.87. PMID 18025970
- [Background] Terrio H, Brenner LA, Ivins BJ, Cho JM, Helmick K, Schwab K, Scally K, Bretthauer R, Warden D. Traumatic brain injury screening: preliminary findings in a US Army Brigade Combat Team. J Head Trauma Rehabil. 2009 Jan-Feb;24(1):14-23. doi: 10.1097/HTR.0b013e31819581d8. PMID 19158592
- [Background] Report to Congress on Mild Traumatic Brain Injury in the United States: Steps to Prevent a Serious Public Health Problem, N.C.f.I.P.a. Control, Editor 2003, Center for Disease Control Prevention: Atlanta, GA.
- [Background] Binder LM, Rohling ML, Larrabee GJ. A review of mild head trauma. Part I: Meta-analytic review of neuropsychological studies. J Clin Exp Neuropsychol. 1997 Jun;19(3):421-31. doi: 10.1080/01688639708403870. PMID 9268816
- [Background] Zakzanis, K.K., L. Leach, and E. Kaplan, Neuropsychological differential diagnosis1999: Swets & Zeitlinger Publishers.
- [Background] Belanger HG, Curtiss G, Demery JA, Lebowitz BK, Vanderploeg RD. Factors moderating neuropsychological outcomes following mild traumatic brain injury: a meta-analysis. J Int Neuropsychol Soc. 2005 May;11(3):215-27. doi: 10.1017/S1355617705050277. PMID 15892898
- [Background] Belanger HG, Vanderploeg RD. The neuropsychological impact of sports-related concussion: a meta-analysis. J Int Neuropsychol Soc. 2005 Jul;11(4):345-57. doi: 10.1017/s1355617705050411. PMID 16209414
- [Background] Tsaousides, T. and W.A. Gordon, Neuropsychological interventions following traumatic brain injury, in Traumatic Brain Injury: Rehabilitative Treatment and Case Management, M.J. Ashley, Editor 2010, CRC Press: Boca Raton, FL.
- [Background] Sohlberg MM, Mateer CA. Improving attention and managing attentional problems. Adapting rehabilitation techniques to adults with ADD. Ann N Y Acad Sci. 2001 Jun;931:359-75. PMID 11462753
- [Background] Sohlberg, M.M. and C.A. Mateer, Attention Process Training-3 (APT-3): A Direct Attention Training Program for the Remediation of the Attention Deficits: APT-3 Manual, 2010, Lash & Associates Publishing/Training Inc.: Youngsville, North Carolina.
- [Background] Ben-Yishay, Y., E.B. Piasetsky, and J. Rattok, A systematic method for ameliorating disorders in basic attention. 1987.
- [Background] Fasotti, L., et al., Time pressure management as a compensatory strategy training after closed head injury. Neuropsychological Rehabilitation, 2000. 10(1): p. 47-65.
- [Background] Sinotte MP, Coelho CA. Attention training for reading impairment in mild aphasia: a follow-up study. NeuroRehabilitation. 2007;22(4):303-10. PMID 17971621
- [Background] Tiersky LA, Anselmi V, Johnston MV, Kurtyka J, Roosen E, Schwartz T, Deluca J. A trial of neuropsychologic rehabilitation in mild-spectrum traumatic brain injury. Arch Phys Med Rehabil. 2005 Aug;86(8):1565-74. doi: 10.1016/j.apmr.2005.03.013. PMID 16084809
- [Background] Cicerone KD. Remediation of "working attention" in mild traumatic brain injury. Brain Inj. 2002 Mar;16(3):185-95. doi: 10.1080/02699050110103959. PMID 11874612
- [Background] Palmese CA, Raskin SA. The rehabilitation of attention in individuals with mild traumatic brain injury, using the APT-II programme. Brain Inj. 2000 Jun;14(6):535-48. doi: 10.1080/026990500120448. PMID 10887887
- [Background] Fahle M. Perceptual learning: specificity versus generalization. Curr Opin Neurobiol. 2005 Apr;15(2):154-60. doi: 10.1016/j.conb.2005.03.010. PMID 15831396
- [Background] Fiorentini A, Berardi N. Perceptual learning specific for orientation and spatial frequency. Nature. 1980 Sep 4;287(5777):43-4. doi: 10.1038/287043a0. PMID 7412873
- [Background] Karni A, Sagi D. Where practice makes perfect in texture discrimination: evidence for primary visual cortex plasticity. Proc Natl Acad Sci U S A. 1991 Jun 1;88(11):4966-70. doi: 10.1073/pnas.88.11.4966. PMID 2052578
- [Background] Poggio T, Fahle M, Edelman S. Fast perceptual learning in visual hyperacuity. Science. 1992 May 15;256(5059):1018-21. doi: 10.1126/science.1589770.
- [Background] Seitz AR, Kim D, Watanabe T. Rewards evoke learning of unconsciously processed visual stimuli in adult humans. Neuron. 2009 Mar 12;61(5):700-7. doi: 10.1016/j.neuron.2009.01.016. PMID 19285467
- [Background] Xiao LQ, Zhang JY, Wang R, Klein SA, Levi DM, Yu C. Complete transfer of perceptual learning across retinal locations enabled by double training. Curr Biol. 2008 Dec 23;18(24):1922-6. doi: 10.1016/j.cub.2008.10.030. Epub 2008 Dec 8. PMID 19062277
- [Background] Hung SC, Seitz AR. Prolonged training at threshold promotes robust retinotopic specificity in perceptual learning. J Neurosci. 2014 Jun 18;34(25):8423-31. doi: 10.1523/JNEUROSCI.0745-14.2014. PMID 24948798
- [Background] Shams L, Seitz AR. Benefits of multisensory learning. Trends Cogn Sci. 2008 Nov;12(11):411-7. doi: 10.1016/j.tics.2008.07.006. PMID 18805039
- [Background] Shibata K, Yamagishi N, Ishii S, Kawato M. Boosting perceptual learning by fake feedback. Vision Res. 2009 Oct;49(21):2574-85. doi: 10.1016/j.visres.2009.06.009. Epub 2009 Jun 14. PMID 19531366
- [Background] Ahissar M, Hochstein S. Task difficulty and the specificity of perceptual learning. Nature. 1997 May 22;387(6631):401-6. doi: 10.1038/387401a0. PMID 9163425
- [Background] Seitz AR, Watanabe T. The phenomenon of task-irrelevant perceptual learning. Vision Res. 2009 Oct;49(21):2604-10. doi: 10.1016/j.visres.2009.08.003. Epub 2009 Aug 7. PMID 19665471
- [Background] Zhang JY, Zhang GL, Xiao LQ, Klein SA, Levi DM, Yu C. Rule-based learning explains visual perceptual learning and its specificity and transfer. J Neurosci. 2010 Sep 15;30(37):12323-8. doi: 10.1523/JNEUROSCI.0704-10.2010. PMID 20844128
- [Background] Green CS, Bavelier D. Action video game modifies visual selective attention. Nature. 2003 May 29;423(6939):534-7. doi: 10.1038/nature01647. PMID 12774121
- [Background] Li R, Polat U, Makous W, Bavelier D. Enhancing the contrast sensitivity function through action video game training. Nat Neurosci. 2009 May;12(5):549-51. doi: 10.1038/nn.2296. Epub 2009 Mar 29. PMID 19330003
- [Background] Deveau J, Lovcik G, Seitz AR. Broad-based visual benefits from training with an integrated perceptual-learning video game. Vision Res. 2014 Jun;99:134-40. doi: 10.1016/j.visres.2013.12.015. Epub 2014 Jan 6. PMID 24406157
- [Background] Klingberg T, Fernell E, Olesen PJ, Johnson M, Gustafsson P, Dahlstrom K, Gillberg CG, Forssberg H, Westerberg H. Computerized training of working memory in children with ADHD--a randomized, controlled trial. J Am Acad Child Adolesc Psychiatry. 2005 Feb;44(2):177-86. doi: 10.1097/00004583-200502000-00010. PMID 15689731
- [Background] Jaeggi SM, Buschkuehl M, Jonides J, Perrig WJ. Improving fluid intelligence with training on working memory. Proc Natl Acad Sci U S A. 2008 May 13;105(19):6829-33. doi: 10.1073/pnas.0801268105. Epub 2008 Apr 28. PMID 18443283
- [Background] Jaeggi SM, Buschkuehl M, Jonides J, Shah P. Short- and long-term benefits of cognitive training. Proc Natl Acad Sci U S A. 2011 Jun 21;108(25):10081-6. doi: 10.1073/pnas.1103228108. Epub 2011 Jun 13. PMID 21670271
- [Background] Klingberg T, Forssberg H, Westerberg H. Training of working memory in children with ADHD. J Clin Exp Neuropsychol. 2002 Sep;24(6):781-91. doi: 10.1076/jcen.24.6.781.8395. PMID 12424652
- [Background] Smith GE, Housen P, Yaffe K, Ruff R, Kennison RF, Mahncke HW, Zelinski EM. A cognitive training program based on principles of brain plasticity: results from the Improvement in Memory with Plasticity-based Adaptive Cognitive Training (IMPACT) study. J Am Geriatr Soc. 2009 Apr;57(4):594-603. doi: 10.1111/j.1532-5415.2008.02167.x. Epub 2009 Feb 9. PMID 19220558
- [Background] Stepankova H, Lukavsky J, Buschkuehl M, Kopecek M, Ripova D, Jaeggi SM. The malleability of working memory and visuospatial skills: a randomized controlled study in older adults. Dev Psychol. 2014 Apr;50(4):1049-1059. doi: 10.1037/a0034913. Epub 2013 Nov 11. PMID 24219314
- [Background] Lilienthal L, Tamez E, Shelton JT, Myerson J, Hale S. Dual n-back training increases the capacity of the focus of attention. Psychon Bull Rev. 2013 Feb;20(1):135-41. doi: 10.3758/s13423-012-0335-6. PMID 23184506
- [Background] Rudebeck SR, Bor D, Ormond A, O'Reilly JX, Lee AC. A potential spatial working memory training task to improve both episodic memory and fluid intelligence. PLoS One. 2012;7(11):e50431. doi: 10.1371/journal.pone.0050431. Epub 2012 Nov 28. PMID 23209740
- [Background] Stephenson, C.L. and D.F. Halpern, Improved matrix reasoning is limited to training on tasks with a visuospatial component. Intelligence, 2013. 41(5): p. 341-357.
- [Background] Kundu B, Sutterer DW, Emrich SM, Postle BR. Strengthened effective connectivity underlies transfer of working memory training to tests of short-term memory and attention. J Neurosci. 2013 May 15;33(20):8705-15. doi: 10.1523/JNEUROSCI.5565-12.2013. PMID 23678114
- [Background] Takeuchi H, Sekiguchi A, Taki Y, Yokoyama S, Yomogida Y, Komuro N, Yamanouchi T, Suzuki S, Kawashima R. Training of working memory impacts structural connectivity. J Neurosci. 2010 Mar 3;30(9):3297-303. doi: 10.1523/JNEUROSCI.4611-09.2010. PMID 20203189
- [Background] Schneiders JA, Opitz B, Krick CM, Mecklinger A. Separating intra-modal and across-modal training effects in visual working memory: an fMRI investigation. Cereb Cortex. 2011 Nov;21(11):2555-64. doi: 10.1093/cercor/bhr037. Epub 2011 Apr 6. PMID 21471559
- [Background] Green CS, Pouget A, Bavelier D. Improved probabilistic inference as a general learning mechanism with action video games. Curr Biol. 2010 Sep 14;20(17):1573-9. doi: 10.1016/j.cub.2010.07.040. PMID 20833324
- [Background] Green CS, Bavelier D. Action-video-game experience alters the spatial resolution of vision. Psychol Sci. 2007 Jan;18(1):88-94. doi: 10.1111/j.1467-9280.2007.01853.x. PMID 17362383
- [Background] Franceschini S, Gori S, Ruffino M, Viola S, Molteni M, Facoetti A. Action video games make dyslexic children read better. Curr Biol. 2013 Mar 18;23(6):462-6. doi: 10.1016/j.cub.2013.01.044. Epub 2013 Feb 28. PMID 23453956
- [Background] Mullins, L., et al., Video tracking of cancellation is sensitive to acute brain impairment and disability. Neurology, 2014. 82(P3): p. 226.
- [Background] Deveau J, Jaeggi SM, Zordan V, Phung C, Seitz AR. How to build better memory training games. Front Syst Neurosci. 2015 Jan 9;8:243. doi: 10.3389/fnsys.2014.00243. eCollection 2014. PMID 25620916
- [Background] Deveau J, Seitz AR. Applying perceptual learning to achieve practical changes in vision. Front Psychol. 2014 Oct 16;5:1166. doi: 10.3389/fpsyg.2014.01166. eCollection 2014. PMID 25360128
- [Background] Bailie, J.M., et al., Neurobehavioral and Cognitive Impact of Mild Traumatic Brain injury: Potential Recruitment Bias, in 33rd Annual Meeting of the National Academy of Neuropsychology 2013, Archives of Clinical Neuropsychology: San Diego, CA.
- [Background] Lange RT, Brickell TA, Kennedy JE, Bailie JM, Sills C, Asmussen S, Amador R, Dilay A, Ivins B, French LM. Factors influencing postconcussion and posttraumatic stress symptom reporting following military-related concurrent polytrauma and traumatic brain injury. Arch Clin Neuropsychol. 2014 Jun;29(4):329-47. doi: 10.1093/arclin/acu013. Epub 2014 Apr 9. PMID 24723461
- [Background] Campbell, J.S., J.H. Greenberg, and J.M. Weil, Confronting mild-TBI and co-occuring PTSD symptoms in combat deployed service members, in Traumatic Brain Injury: A Neurologic Approach to Diagnosis, Management, and Rehabilitation, J.W. Tsao, Editor 2012, Springer Press: New Yor, NY.
- [Background] Campbell, J.S., et al., Evaluation of Post-deployment Screening for Traumatic Brain Injury and Blast Exposure in a Sample of High-Risk Sailors Deployed to Iraq, in Coping with Blast-Related Traumatic Brain injury in Returning Troops2011, IOS Press: Washington, DC. p. 126-128.
- [Background] Malec, J.F., Goal attainment scaling in rehabilitation. Neuropsychological Rehabilitation, 1999. 9(3-4): p. 253-275.
- [Background] Rabin LA, Barr WB, Burton LA. Assessment practices of clinical neuropsychologists in the United States and Canada: a survey of INS, NAN, and APA Division 40 members. Arch Clin Neuropsychol. 2005 Jan;20(1):33-65. doi: 10.1016/j.acn.2004.02.005. PMID 15620813
- [Background] Bogner J, Corrigan JD. Reliability and predictive validity of the Ohio State University TBI identification method with prisoners. J Head Trauma Rehabil. 2009 Jul-Aug;24(4):279-91. doi: 10.1097/HTR.0b013e3181a66356. PMID 19625867
- [Background] Corrigan JD, Bogner J. Initial reliability and validity of the Ohio State University TBI Identification Method. J Head Trauma Rehabil. 2007 Nov-Dec;22(6):318-29. doi: 10.1097/01.HTR.0000300227.67748.77. PMID 18025964
- [Background] Whitney KA, Shepard PH, Mariner J, Mossbarger B, Herman SM. Validity of the Wechsler Test of Adult Reading (WTAR): effort considered in a clinical sample of U.S. military veterans. Appl Neuropsychol. 2010 Jul;17(3):196-204. doi: 10.1080/09084282.2010.499787. PMID 20799111
- [Background] Stern, R.A. and T. White, Neuropsychological Assessment Battery: Administration, scoring, and interpretation manual, 2003, Psychological Assessment Resources: Lutz, FL.
- [Background] Stern, R.A. and T. White, NAB Naming Test: Professional Manual, 2009, Psychological Assessment Resources: Lutz, FL.
- [Background] Homack S, Riccio CA. Conners' Continuous Performance Test (2nd ed.; CCPT-II). J Atten Disord. 2006 Feb;9(3):556-8. doi: 10.1177/1087054705283578. No abstract available. PMID 16481673
- [Background] Smith, A., Symbol Digits Modalities Test: Manual, 2007, Western Psychological Services: Los Angeles.
- [Background] Weathers, F.W., J.A. Huska, and T.M. Keane, PTSD Checklist- Military Version (PCLM), 1991, National Center for PTSD- Behavioral Science Division.
- [Background] Gewirtz AH, Polusny MA, DeGarmo DS, Khaylis A, Erbes CR. Posttraumatic stress symptoms among National Guard soldiers deployed to Iraq: associations with parenting behaviors and couple adjustment. J Consult Clin Psychol. 2010 Oct;78(5):599-610. doi: 10.1037/a0020571. PMID 20873896
- [Background] Cook JM, Elhai JD, Cassidy EL, Ruzek JI, Ram GD, Sheikh JI. Assessment of trauma exposure and post-traumatic stress in long-term care veterans: preliminary data on psychometrics and post-traumatic stress disorder prevalence. Mil Med. 2005 Oct;170(10):862-6. doi: 10.7205/milmed.170.10.862. PMID 16435760
- [Background] Belanger HG, Kretzmer T, Vanderploeg RD, French LM. Symptom complaints following combat-related traumatic brain injury: relationship to traumatic brain injury severity and posttraumatic stress disorder. J Int Neuropsychol Soc. 2010 Jan;16(1):194-9. doi: 10.1017/S1355617709990841. Epub 2009 Sep 17. PMID 19758488
- [Background] Polusny MA, Kehle SM, Nelson NW, Erbes CR, Arbisi PA, Thuras P. Longitudinal effects of mild traumatic brain injury and posttraumatic stress disorder comorbidity on postdeployment outcomes in national guard soldiers deployed to Iraq. Arch Gen Psychiatry. 2011 Jan;68(1):79-89. doi: 10.1001/archgenpsychiatry.2010.172. PMID 21199967
- [Background] van Veldhoven LM, Sander AM, Struchen MA, Sherer M, Clark AN, Hudnall GE, Hannay HJ. Predictive ability of preinjury stressful life events and post-traumatic stress symptoms for outcomes following mild traumatic brain injury: analysis in a prospective emergency room sample. J Neurol Neurosurg Psychiatry. 2011 Jul;82(7):782-7. doi: 10.1136/jnnp.2010.228254. Epub 2011 Jan 17. PMID 21242288
- [Background] Using the PTSD checklist U.S. Department of Veterans Affairs, V.N.C.f. PTSD, Editor 2012.
- [Background] Bliese PD, Wright KM, Adler AB, Cabrera O, Castro CA, Hoge CW. Validating the primary care posttraumatic stress disorder screen and the posttraumatic stress disorder checklist with soldiers returning from combat. J Consult Clin Psychol. 2008 Apr;76(2):272-81. doi: 10.1037/0022-006X.76.2.272. PMID 18377123
- [Background] Yeager DE, Magruder KM, Knapp RG, Nicholas JS, Frueh BC. Performance characteristics of the posttraumatic stress disorder checklist and SPAN in Veterans Affairs primary care settings. Gen Hosp Psychiatry. 2007 Jul-Aug;29(4):294-301. doi: 10.1016/j.genhosppsych.2007.03.004. PMID 17591505
- [Background] Kroenke K, Spitzer RL, Williams JB. The PHQ-9: validity of a brief depression severity measure. J Gen Intern Med. 2001 Sep;16(9):606-13. doi: 10.1046/j.1525-1497.2001.016009606.x. PMID 11556941
- [Background] Lowe B, Spitzer RL, Grafe K, Kroenke K, Quenter A, Zipfel S, Buchholz C, Witte S, Herzog W. Comparative validity of three screening questionnaires for DSM-IV depressive disorders and physicians' diagnoses. J Affect Disord. 2004 Feb;78(2):131-40. doi: 10.1016/s0165-0327(02)00237-9. PMID 14706723
- [Background] Spitzer RL, Kroenke K, Williams JB. Validation and utility of a self-report version of PRIME-MD: the PHQ primary care study. Primary Care Evaluation of Mental Disorders. Patient Health Questionnaire. JAMA. 1999 Nov 10;282(18):1737-44. doi: 10.1001/jama.282.18.1737. PMID 10568646
- [Background] Williams JW Jr, Noel PH, Cordes JA, Ramirez G, Pignone M. Is this patient clinically depressed? JAMA. 2002 Mar 6;287(9):1160-70. doi: 10.1001/jama.287.9.1160. PMID 11879114
- [Background] Fann JR, Bombardier CH, Dikmen S, Esselman P, Warms CA, Pelzer E, Rau H, Temkin N. Validity of the Patient Health Questionnaire-9 in assessing depression following traumatic brain injury. J Head Trauma Rehabil. 2005 Nov-Dec;20(6):501-11. doi: 10.1097/00001199-200511000-00003. PMID 16304487
- [Background] Gronwall DM. Paced auditory serial-addition task: a measure of recovery from concussion. Percept Mot Skills. 1977 Apr;44(2):367-73. doi: 10.2466/pms.1977.44.2.367. PMID 866038
- [Background] Kolitz BP, Vanderploeg RD, Curtiss G. Development of the Key Behaviors Change Inventory: a traumatic brain injury behavioral outcome assessment instrument. Arch Phys Med Rehabil. 2003 Feb;84(2):277-84. doi: 10.1053/apmr.2003.50100. PMID 12601661